CLINICAL TRIAL: NCT05119803
Title: Investigation of the Relationship of Spinal Alignment and Spinal Mobility on Upper Extremity Functions and Quality of Life in Patients With Parkinson's Disease.
Brief Title: The Relationship of Spine Posture and Mobility With Upper Extremity Functions in Parkinson's Patients
Status: Completed | Type: Observational
Sponsor: Gulhane School of Medicine (Other)
Responsible Party: Principal Investigator, Mustafa Ertuğrul Yaşa, Assoc. Prof, Gulhane School of Medicine
Other Study IDs: 2021-335
Record Dates: First submitted 2021-11-03; First posted 2021-11-15 (Actual); Last update posted 2022-07-08 (Actual); Status verified 2022-07

CONDITIONS: Parkinson; Posture; Upper Extremity; Quality of Life
Keywords: Parkinson; Posture; Upper Extremity; Quality of Life; Spinal Curvatures
MeSH Terms: conditions — Spinal Curvatures

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Parkinson's patients: The cognitive status of the participants will be evaluated using the 'Standardized Mini Mental Test'.
  The 'Unified Parkinson's Disease Assessment Scale Part 3' will be used to evaluate the motor function of Parkinson's patients.
  Spinal posture will be assessed using the IDIAG M360 (IDIAG, Fehraltorf, Switzerland) Spinal Mouse. This device is an electronic computer aided measuring device that measures the range of motion of the spine and evaluates the angle and shape of the spine in the sagittal and frontal planes.
  The upper extremity functions of Parkinson's patients will be evaluated with the '9-Hole Peg Test'.
  A short version of PDQ-39, called the 8-item Parkinson's Disease Questionnaire (PDQ-8), will be applied to determine the quality of life of Parkinson's patients. The PDQ-8 consists of eight items that belong to each of the eight dimensions in the original PDQ-39.
  Interventions: Device: Spinal Mouse (IDIAG M360 ); Other: Nine Hole Peg Test
- Healthy control group: The cognitive status of the participants will be evaluated using the 'Standardized Mini Mental Test'. This scale is frequently used for the general determination of the cognitive status of individuals rather than for the purpose of diagnosis.
  The upper extremity functions of healty control group will be evaluated with the '9-Hole Peg Test'.
  Spinal posture will be assessed using the IDIAG M360 (IDIAG, Fehraltorf, Switzerland) Spinal Mouse. This device is an electronic computer aided measuring device that measures the range of motion of the spine and evaluates the angle and shape of the spine in the sagittal and frontal planes.
  Interventions: Device: Spinal Mouse (IDIAG M360 ); Other: Nine Hole Peg Test

INTERVENTIONS:
Device: Spinal Mouse (IDIAG M360 ) — This device is an electronic computer-aided measuring december that measures the range of motion of the spine, evaluates the angle and shape of the spine in the sagittal and frontal planes. The device provides data to the computer via Bluetooth, and the measured curvatures are displayed on the computer screen. The method has no medical risks or dangers. The device has two rotating wheels that follow the spinous protrusions of the spine, and the distance and angle measurements are transferred from the device to the computer.
Other: Nine Hole Peg Test — The nine-hole peg test is a simple, fast and manual skill test that has been proven to be valid and reliable in measuring upper limb function in Parkinson's patients. While the patient is sitting, he is asked to insert nine sticks into the holes of the test box with nine holes one by one as fast as possible and remove them back when he is finished

SUMMARY:
The aim of this study is to investigate whether spinal alignment and spinal mobility have an effect on upper extremity functions in Parkinson's patients. In the light of the data obtained as a result, we think that our study will also contribute to determining the factors that may cause upper limb dysfunctions seen in Parkinson's patients and will guide new treatment-oriented studies to be carried out in the future.

DETAILED DESCRIPTION:
Parkinson's disease is a neurodegenerative disease that occurs due to the influence of dopaminergic pathways, causing progressive deficits, especially in motor functions. The four main motor symptoms of Parkinson's are tremor, muscular rigidity, bradykinesia (slowing down of movements) and postural instability.

One of the inadequacies of these symptoms on patients is the disruption of the functions of the upper extremities. Since the formation of isometric force at parkinson disease is delayed, the reaction time is disrupted. In addition, patients exhibit sensory deficits, such as a decrease in the spatial and temporal tactile discrimination thresholds of the fingertips. Since patients tend to have difficulty initiating movement to a goal (akinesia), there are disorders of reaching and grasping it. There is also a lack of coordination between the timing of the movement components. In particular, tremor and rigidity can cause serious deficiencies during targeted activities in which the patient uses their upper limbs in their daily life. Incidence studies conducted to date have shown that Parkinson disease, causes various degrees of impairment in the manual skills of about 90% of individuals. In this context, the fine manipulative skills of the hand and the identification of components affecting the functions of the upper extremities in this group of diseases are important in the detection and management of the problem.

In Parkinson's disease, forward oblique posture, forward tilting of the head and neck, and scoliosis are common spinal deformities. The studies conducted have revealed that these deformities are directly proportional to the severity of the disease. In addition, the rigidity of the global trunk muscles may reduce the spinal mobility of the patients and may affect the independence measures in trunk-dependent activities. In this regard, it is important to analyze the spine sequence and mobility when monitoring patients in this group of diseases. At the same time, postural correction and balance reactions are also reduced due to postural changes, such as the development of flexion posture and reduced body rotation in Parkinson's disease. This condition causes Parkinson's patients to have difficulty maintaining their current posture and an increased risk of falling.

In a study conducted with healthy adults, upper extremity function was evaluated using the 'Jebsen Taylor Hand Function Test' in three different trunk postures (flexion, lateral flexion, neutral posture), and the best upper limb performance was obtained in neutral trunk posture. In another study, it was found that Pisa Syndrome (lateral flexion deformity of the trunk) was associated with both upper extremity functions and the level of independence in activities of daily living in Parkinson's disease. To the best of our group's knowledge, extremity dysfunctions, spinal posture and mobility involvement in Parkinson's disease have been well defined in the studies we have conducted in the literature, but we have not found any study investigating the effects of spinal alignment and spinal mobility on upper extremity functions and quality of life.

The aim of this study, which was planned accordingly, was to investigate: (A) spinal postural changes in Parkinson's disease, (B) changes in upper extremity functions in Parkinson's disease, (C) effects of spinal alignment and spinal mobility on upper extremity functions and quality of life in Parkinson's disease.

ELIGIBILITY:
Inclusion Criteria:

For Parkinson's Patients;

* Being 18 years or older
* Receiving a diagnosis of Parkinson's made by a specialist neurologist
* Being able to walk independently
* Being between stages 1-4 on the Hoehn & Yahr scale

For the Control Group;

• Being 18 years or older

Exclusion Criteria:

For Parkinson's Patients;

* Having any neurological disease other than Parkinson's
* Presence of cardiovascular, vestibular and musculoskeletal disease
* Having a score of <24 on the Standardized Mini Mental Test

For the Control Group;

* Having any disease that may affect balance, gait, posture and respiratory functions
* Using sedative - antidepressant medication that will impair physical well-being
* Having a score of <24 on the Standardized Mini Mental Test

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy individuals with similar age and body mass index values for Parkinson's patients who were diagnosed with Parkinson's disease according to the UK Parkinson's Disease Association Brain Bank criteria, followed in the Health Sciences University Gülhane Training and Research Hospital Neurology Department Parkinson's Polyclinic, and the control group will be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2021-11-03 (Actual); Primary Completion 2022-02-03 (Actual); Study Completion 2022-06-15 (Actual)

PRIMARY OUTCOMES:
Spinal Mouse | Measurements will begin on the estimated 3 November and will end on the estimated June 2022.
  This device is an electronic computer aided measuring device that measures the range of motion of the spine and evaluates the angle and shape of the spine in the sagittal and frontal planes. The device provides data to the computer via Bluetooth and the measured curvatures are displayed on the computer screen. The method has no medical risk or danger. The device has two rotating wheels that follow the spinous processes of the spine and the distance and angle measurements are transferred from the device to the computer. This information is then used to calculate the relative positions of each vertebra, the angles between the vertebrae, and the total angle of the frontal and sagittal plane curvatures with its software.

SECONDARY OUTCOMES:
Nine Hole Peg Test | Measurements will begin on the estimated 3 November and will end on the estimated June 2022.
  It is a simple, fast, manual skill test with proven validity and reliability. It is particularly sensitive to changes in upper extremity performance. The test material consists of nine small sticks made in standard sizes and a nine-hole board on which to place them. In the test, while the patient is in a sitting position, the patient is asked to line up the 9 sticks inside the box on the table as quickly as possible into the holes of the other box and immediately remove it after finishing. The test is started with the dominant hand. The time elapsed between the moment the hand touches the bars and the placing of the last bar in the box is recorded as the result of the test.

OTHER OUTCOMES:
Parkinson's Disease Questionnaire (PDQ-8) | Measurements will begin on the estimated 3 November and will end on the estimated June 2022.
  In order to determine the quality of life of Parkinson's patients, the short version of the PDQ-39, called the 8-item Parkinson's Disease Questionnaire (PDQ-8) will be administered. The PDQ-8 consists of eight items belonging to each of the eight dimensions in the original PDQ-39.
  The PDQ-8 has some advantages over the PDQ-39 such as being easier to use, more practical and less time consuming.

CONTACTS AND LOCATIONS:
Locations (1):
- Sağlık Bilimleri Üniversitesi, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No